CLINICAL TRIAL: NCT03761706
Title: Impact of Home-based Aerobic and Strength Exercises During Chemotherapy for Early Breast Cancer on Biomarkers of Aging and Patient-reported Symptoms and Outcomes
Brief Title: Impact of Home-based Aerobic and Strength Exercises During Chemotherapy for Early Breast Cancer on Biomarkers of Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Breast Cancer Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LCCC 1749
Record Dates: First submitted 2018-06-05; First posted 2018-12-03 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: breast cancer; exercise; chemotherapy and aging
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Cohort (Experimental): This is a one-arm intervention study that includes assessments and questionnaires at several time points as early stage breast cancer patients undergo chemotherapy and at 6 months post-chemotherapy. Study participants will be asked to wear a FitBit provided by the research team and agree to FitBit data downloads during regularly scheduled chemotherapy clinic visits to evaluate engagement in physical activity. Study participants will complete questionnaires, an exercise log, and submit blood samples as multiple time points.
  Interventions: Behavioral: Engagement in Physical Activity; Other: Questionnaires

INTERVENTIONS:
Behavioral: Engagement in Physical Activity — Study participants will be asked to wear a FitBit provided by the research team and agree to FitBit data downloads during regularly scheduled chemotherapy clinic visits. Participants will also complete a daily exercise log to record the total number of minutes walked and the total number of steps from the FitBit.
Other: Questionnaires — Study participants will complete the following questionnaires: Health Behavior Questionnaire (HBQ), Short Physical Performance Battery (SPPB), Functional Assessment of Cancer Therapy-General (FACT-G), 4.4.5 Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F), PROMIS Cognitive Function (Short Form 8a), Functional Assessment of Cancer-Gynecology Oncology Group-Neurotoxicity (FACT/GOG-NTX-12) Version 4, Nutrition Survey, Perceived Self-Efficacy for Fatigue Self-Management (PSEFSM),

SUMMARY:
Purpose: To determine if engagement in physical activity during chemotherapy will have a moderating effect on increases in p16 levels during chemotherapy.

Participants: 200 patients age 21 or older with a Stage I-III breast cancer diagnosis who are about to start adjuvant or neoadjuvant chemotherapy.

Procedures: The study entails screening, recruiting and consenting 200 eligible breast cancer patients who are about to begin adjuvant or neoadjuvant chemotherapy and agree to participate in a physical activity intervention, maintain a printed daily exercise log, wear a FitBit, complete questionnaires and assessments, and provide blood samples at various time points.

DETAILED DESCRIPTION:
The overall focus of this study remains the investigation of associations between p16 and assessments (independent and patient-reported) of chemotherapy-related toxicity (adverse events and symptoms) and patient-reported measures of function and quality of life. The research team has determined that p16 increases dramatically during chemotherapy and that p16 levels among persons of similar age are lower among those who exercise as compared to those who are sedentary. The research team hypothesizes that engagement in physical activity during chemotherapy will have a moderating effect on increases in p16 levels during chemotherapy. To test this hypothesis, the study proposes to build on a completed trial, LCCC1334, and enroll 200 evaluable patients age 21-64 with a Stage I-III breast cancer diagnosis who are about to start adjuvant or neoadjuvant chemotherapy in an intervention that entails both aerobic and resistance exercises.

Results from both LCCC1334 and LCCC1410 and the proposed study, LCCC1749, will be used to provide evidence for a future grant application to conduct a randomized controlled trial in a larger study population to (1) establish the effect of physical activity on p16 levels during chemotherapy and (2) further evaluate how baseline and post-chemotherapy p16 levels correlate with measures of treatment-related toxicity and patient-reported outcomes over time. Findings from this study will also provide preliminary evidence for further investigations of the potential benefits of exercise during early breast cancer chemotherapy for (1) reducing the incidence and severity of peripheral neuropathy and (2) managing the interface of fatigue and perceived cognition deficits.

ELIGIBILITY:
Inclusion Criteria:

* Study subjects must meet all of the inclusion criteria listed below to participate in this study:
* 21 years of age or older, female
* Histologically confirmed Stage I, II or III breast cancer (if the patient has had more than one breast cancer, then the most recent diagnosis)
* Scheduled to begin an appropriate adjuvant or neo-adjuvant chemotherapy regimen as defined by NCCN guidelines (www.nccn.org). Patients receiving anti-HER-2 therapy are eligible but the intervention will only be tested during the chemotherapy portion of the regimen.
* English speaking
* IRB approved, signed written informed consent
* Approval from their treating physician to engage in moderate-intensity physical activity
* Patient-assessed ability to walk and engage in moderate physical activity
* Willing and able to meet all study requirements.

Exclusion Criteria:

* All subjects meeting any of the exclusion criteria at baseline will be excluded from study participation. Exclusion criteria are:
* One or more significant medical conditions that in the physician's judgment preclude participation in the walking or strength training intervention.
* Unable to walk or engage in moderate-intensity physical activity.

Ages: 21 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 132 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Compare the change in p16 from baseline to end of chemotherapy | Baseline, 6-months post Baseline, 12-months post-Baseline
  Compare the change in p16 from baseline to end of chemotherapy for patients receiving a physical activity intervention to the historical value seen in previous studies (LCCC810 and 1027) of similar patients who did not participate in a physical activity intervention.

SECONDARY OUTCOMES:
Measure association of physical activity levels (Fitbit steps and strength training) with change in p16 levels | Baseline, during Chemotherapy (from 1st infusion through last infusion, which varies widely by chemotherapy regimen -- from 12 weeks to 30 weeks) , and 12-months post-Baseline
  Will upload Fitbit and collect strength training data to evaluate the association of physical activity levels (Fitbit steps) with change in p16 levels.
Measure associations between weight, physical activity and diet during chemotherapy. | Baseline, 3-months post-Baseline, 6-months post-Baseline, and 12-months post-Baseline
  Will administer the NHANES Nutrition Survey at several time points during the study. The NHANES survey is not a scale. It is not scored. It is descriptive, asking about the frequency of consumption of specific items.
Chemotherapy-induced peripheral neuropathy (CIPN) as assessed by the FACT/GOG-NTX | Baseline, During Chemotherapy (from 1st infusion through last infusion, which varies widely by chemotherapy regimen -- from 12 weeks to 30 weeks), 6-months post Baseline, 12-months post-Baseline
  Will administer the FACT/GOG-NTX instrument.
Chemotherapy-induced peripheral neuropathy (CIPN) as assessed by the CTCAE. | Baseline, During Chemotherapy (from 1st infusion through last infusion, which varies widely by chemotherapy regimen -- from 12 weeks to 30 weeks), 6-months post Baseline, 12-months post-Baseline
  Will administer the CTCAE.
Chemotherapy-induced peripheral neuropathy (CIPN) as assessed by the PRO-CTCAE. | Baseline, During Chemotherapy (from 1st infusion through last infusion, which varies widely by chemotherapy regimen -- from 12 weeks to 30 weeks), 6-months post Baseline, 12-months post-Baseline
  Will administer the PRO-CTCAE.
Chemotherapy-induced peripheral neuropathy (CIPN) as assessed by the SPPB. | Baseline, During Chemotherapy (from 1st infusion through last infusion, which varies widely by chemotherapy regimen -- from 12 weeks to 30 weeks), 6-months post Baseline, 12-months post-Baseline
  Will administer the Short Physical Performance Battery (SPPB).
Measure association of p16 with changes in QOL measures as assessed by the FACT-G | Baseline, 6-months post-Baseline, 12-months post-Baseline
  Will administer the FACT-G Questionnaire. The FACT-G is scored in a Likert-type scale from 0+not at all to 4=very much. Higher scores signify higher quality of life. Subscales are physical, social/family, emotional and functional -- which are analyzed separately and can be combined into a total FACT-G score.
Measure association of p16 with changes in QOL measures as assessed by the FACIT-F | Baseline, 6-months post-Baseline, 12-months post-Baseline
  Will administer the FACIT-F Questionnaire. This Likert-type scale ranges from 0=not at all to 4=very much, with higher scores signifying higher fatigue. No subscales.
Measure association of p16 with changes in QOL measures as assessed by the MHI-17 | Baseline, 6-months post-Baseline, 12-months post-Baseline
  Will administer the MHI-17 Health Questionnaire. This 17 item measure consists of two subscales -- Anxiety and Depression. The Likert-type scale ranges from 0=all of the time to 5=none of the time. Higher scores indicate higher anxiety or depression. The two subscales are not combined into one MHI score.
Measure association of p16 with changes in QOL measures as assessed by the MOS Social Activity Limitation Questionnaire | Baseline, 6-months post-Baseline, 12-months post Baseline
  Administer the MOS Social Activity Limitation Questionnaire. We are using only one item from this scale. Likert-type scoring is 0=all of the time to4=none of the time. Higher score signifies less interference with social activities.
Measure association of p16 with changes in QOL measures as assessed by the PROMIS Instrumental Support | Baseline, 6-months post Baseline, 12-months post-Baseline
  Administer the PROMIS Instrumental Support Questionnaire. This Likert-type scale is from 1=never to 5=always. Higher score signifies higher instrumental support. No subscales.
Measure association of p16 with changes in QOL measures as assessed by the PROMIS Social Isolation Questionnaire. | Baseline, 6-months post-Baseline, 12-months post-Baseline
  Administer PROMIS Social Isolation Questionnaire. Likert-type scoring is 0=never to 5=alwayse. Higher score signifies more social isolation. No subscales.
Measure association of p16 with changes in QOL measures as assessed by the PROMIS Global Health | Baseline, 6-months post-Baseline, 12-months post-Baseline
  Administer PROMIS Global Health Questionnaire. Likert-type scale from 0=excellent to 4=poor. Higher score signifies lower global health. No subscales.
Measure association of p16 with changes in cognition by the PROMIS Cognitive Function-Short Form | Baseline, 6-months post-Baseline
  Will administer the PROMIS Cognitive Function-Short Form (8a). This Likert-type scale is from 1=very often to 5=never. Higher scores signify higher cognitive function. No subscales.
Measure association of p16 with changes in cognition by the Blessed Memory Concentration test (BOMC) | Baseline, 6-months post-Baseline
  Will administer the Blessed Memory Concentration test (BOMC).
Measure association of p16 with changes in functional status by the Timed Up and Go Test | Baseline, 6-months post-Baseline
  Administer theTimed Up and Go Test
Measure association of p16 with changes in functional status by the Medical Outcomes Survey. | Baseline, 6-months post-Baseline
  Administer the Medical Outcomes Survey. Likert-type scale from 0=without help to 2=completely unable. Higher score signifies more limitations. No subscale.
Measure association of p16 with changes in functional status with the Instrumental Activities of Daily Living Survey | Baseline, 6-months post-Baseline
  Administer the Instrumental Activities of Daily Living Survey. This Likelrt-type scale is from 0=without help to 2=completely unable. Higher scores signify greater limitations. No subscale.
Measure association of p16 with changes in functional status with the Karnofsky Performance Status | Baseline, 6-months post-Baseline
  Administer the Karnofsky Performance Status
Measure association of p16 with number of Fall Questionnaire | Baseline, 6-months post-Baseline
  One question will inquire about falls within the past 6 months.
Measure association of p16 with limitations in walking one block | Baseline, 6-months post-Baseline
  One question will inquire whether the participant's health limits their ability to walk one block = range 0=limited a lot to 2=not limited at all

OTHER OUTCOMES:
Measure association of p16 with body composition | Baseline, During Chemotherapy (from 1st infusion through last infusion, which varies widely by chemotherapy regimen -- from 12 weeks to 30 weeks), 6-months post-Baseline and 12-months post-Baseline
  Evaluate the association of p16 with body composition measures (Bioimpedence, DEXA or BMI) at baseline and over time. p16 is the outcome of interest. We will analyze the correlation between p16 and (1) DEXA or (2) BMI or (3) bioimpedence -- BMI will be available for all participants, while DEXA and bioimpedence measures will not necessarily be available for all participants.
Mean change in p16 between baseline to end of chemo, compared to previous studies | Baseline, 6-months post-Baseline
  Mean change in p16 levels measured between baseline to end of chemotherapy, as compared to the historical value seen in previous studies (LCCC810 and 1027) of similar patients who did not participate in a physical activity intervention

CONTACTS AND LOCATIONS:
Overall Officials: Hyman B. Muss, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nyrop KA, Page A, Deal AM, Wagoner C, Kelly EA, Kimmick GG, Copeland A, Speca J, Wood WA, Muss HB. Association of self-directed walking with toxicity moderation during chemotherapy for the treatment of early breast cancer. Support Care Cancer. 2023 Dec 28;32(1):68. doi: 10.1007/s00520-023-08275-4. PMID 38153568